CLINICAL TRIAL: NCT02183168
Title: A Randomized, Open Label, 3-arm Evaluation of Efficacy and Safety of Meloxicam Suppository (15mg Daily) and Tablet (15 mg Daily) Compared to Indomethacin Suppository (50 mg Daily) in Patients With Ankylosing Spondylitis
Brief Title: Evaluation of Efficacy and Safety of Meloxicam Suppository (15mg Daily) and Tablet (15 mg Daily) Compared to Indomethacin Suppository (50 mg Daily) in Patients With Ankylosing Spondylitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 107.237
Record Dates: First submitted 2014-07-04; First posted 2014-07-08 (Estimated); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Spondylitis, Ankylosing
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Meloxicam; Indomethacin

ARMS (3):
- Meloxicam suppository (Experimental)
  Interventions: Drug: Meloxicam suppository
- Meloxicam tablet (Experimental)
  Interventions: Drug: Meloxicam tablet
- Indomethacin suppository (Active Comparator)
  Interventions: Drug: Indomethacin

INTERVENTIONS:
Drug: Meloxicam suppository
  Arms: Meloxicam suppository
Drug: Meloxicam tablet
  Arms: Meloxicam tablet
Drug: Indomethacin
  Arms: Indomethacin suppository

SUMMARY:
Study to assess the efficacy and safety of meloxicam suppository 15 mg once daily, meloxicam tablet 15 mg once daily compared with Indomethacin suppository (50 mg daily) in patients with ankylosing spondylitis

ELIGIBILITY:
Inclusion Criteria:

* Active ankylosing spondylitis (pain rated >= 40 mm on a VAS and increased of at least 30% after nonsteroidal anti-inflammatory drugs (NSAIDs) wash-out)), without peripheral arthritis and inflammatory bowel disease

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2001-07-01 (Actual); Primary Completion 2002-05-01 (Actual)

PRIMARY OUTCOMES:
Overall pain during the previous 48 hours assessed on a Visual Analogue Scale (VAS) | 6 weeks
Functional Index of ankylosing spondylitis of Dougados | 6 weeks
Overall assessment of disease activity by the patient on VAS | 6 weeks

SECONDARY OUTCOMES:
Overall assessment of disease activity by the investigator on a VAS | 6 weeks
Global efficacy assessed by the patient (verbal rating scale) | 6 weeks
Global efficacy assessed by the investigator (verbal rating scale) | 6 weeks
Duration of morning stiffness | 6 weeks
Evaluation of spinal pain by the investigator (verbal rating scale) | 6 weeks
Assessment of Schober test | 6 weeks
Assessment of Chest expansion | 6 weeks
Assessment of Fingers - to - floor test | 6 weeks
Assessment of Night pain (verbal rating scale) | 6 weeks
Total number of study withdrawals | 6 weeks
Number of study withdrawals due to lack of efficacy | 6 weeks
Assessment of Paracetamol consumption | 6 weeks
Assessment of Patient status with regard to disease condition | 6 weeks